CLINICAL TRIAL: NCT01403883
Title: Impact of Psychological and Enterostomal Therapy Care for Patient Undergoing Rectal Cancer Resection With a Temporary Stoma. Monocentric Randomized Study
Brief Title: Psychological and Enterostomal Therapy Care
Acronym: PROSPER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Association de Recherche Experimentale et Clinique en Chirurgie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: UK10005
Record Dates: First submitted 2010-11-30; First posted 2011-07-27 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2015-01

CONDITIONS: Cancer of Rectum
Keywords: Rectal cancer; Temporary stoma; Psychological disorders
MeSH Terms: conditions — Rectal Neoplasms; Mental Disorders | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (Active Comparator): standard care of patient with psychological and enterostomal therapy clinic if necessary
  Interventions: Behavioral: Standard Care
- Optimal care (Experimental): Optimal care of patient with systematic and repeated psychological and enterostomal therapy follow up
  Interventions: Behavioral: Optimal care (Psychological and enterostomal therapy clinics)

INTERVENTIONS:
Behavioral: Standard Care — Psychological & enterostomal therapy clinics on demand only
  Arms: Standard care
Behavioral: Optimal care (Psychological and enterostomal therapy clinics) — Psychological clinics at D-45, D0, D45, D60, D90 enterostomal therapy clinics at D-45, D0, D45, D60
  Arms: Optimal care

SUMMARY:
In case of rectal cancer surgery, temporary stoma is recommended to decrease the risk of postoperative anastomotic leakage. The aim of the study was to assess the benefit of an optimal care, i.e., both psychological and enterostomal therapy care.

DETAILED DESCRIPTION:
The aim of the study is to asses the benefit of an optimal and specific care concerning the temporary stoma in patients operated for rectal cancer surgery in term of psychological and enterostomal therapy effect.

This study is a monocentric and randomized trial.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 y
* Rectal adenocarcinoma (tumor height < 15 cm from the anal verge) with or without pre operative radiochemotherapy.
* Open or laparoscopic rectal excision with partial or total meso rectal excision with sphincter preservation by colo rectal or colo anal anastomosis.
* Temporary stoma.
* Patient consent
* Patient with national health affiliation

Exclusion Criteria:

* Stage IV disease with synchronous hepatic or pulmonary metastases
* Colonic cancer > 16 cm
* Associated surgical procedure (Hepatic resection, small bowel resection subtotal colectomy)
* Abdominal perineal resection
* Associated comorbidity
* Emergency surgery
* Psychological care refusal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2011-10; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Evolution of Global Quality of life (SF36) | at Day45, Day0, Day45, Day60, Day90
Evolution of Psychological anxiety score (STAI/Beck) | at Day-45, Day0, Day45, Day60, Day90

SECONDARY OUTCOMES:
Evolution of Specific stoma score and stoma care learning | at Day-45, Day0, Day45, Day60, Day90
Hospital stay | at Day90
Overall morbidity | at Day45, Day60, Day90
Specific stoma related morbidity | at Day45, Day60, Day90

CONTACTS AND LOCATIONS:
Overall Officials: Yves PANIS, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France